CLINICAL TRIAL: NCT01225016
Title: Characterization of Thyroid Nodules Using Contrast Enhanced Ultrasound
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funding and issues with ability to complete all procedures, it was decided that this study could not be carried out and therefore withdrawn.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Glenn Peters, MD, Professor of Surgery, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UAB 1007
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Definity contrast agent — Thyroid ultrasound using contrast agent

SUMMARY:
This study will evaluate thyroid nodules using specialized ultrasound imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with a thyroid nodule 2. Age greater than or equal to 19 years of age 3. Patients must sign informed consent

Exclusion Criteria:

* 1. Women who are pregnant or nursing 2. Patients with pulmonary hypertension, unstable cardiopulmonary condition,or right to left shunt 3. Hypersensitivity to perfluten 4. Psychological condition that renders the patient unable to understand the informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To estimate the accuracy (sensitivity and specificity) of the contrast enhanced ultrasound for characterization of thyroid nodules. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Glenn E Peters, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Universith of Alabama at Birmingham, Birmingham, Alabama, United States